CLINICAL TRIAL: NCT00063427
Title: A Phase 2, Open-Label Study of MAC-321 Administered Intravenously as a Single Agent for the Treatment of Advanced Colorectal Cancer
Brief Title: Study Evaluating MAC-321 in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3128K1-200
Record Dates: First submitted 2003-06-26; First posted 2003-06-27 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms
Keywords: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — MAC321

INTERVENTIONS:
Drug: MAC-321

SUMMARY:
Assess the clinical activity of MAC-321 administered IV as a second-line or third-line antineoplastic agent to subjects with advanced colorectal cancer. Clinical activity will be assessed by determining the percentage of subjects exhibiting an objective response (complete plus partial responses). Tumor response will be assessed following modified Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histologic and/or cytologic diagnosis of metastatic or relapsed colorectal cancer at any time during disease but not candidates for surgical resection.
* Prior treatment with at least 1 conventional approved therapeutic regimen.
* Subjects who have failed prior cytotoxic chemotherapy regimens containing irinotecan (CPT-11), 5 fluorouracil (5-FU), and/or oxaliplatin for advanced (relapsed) metastatic colon cancer are eligible

Exclusion Criteria:

* Other chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks before signing the ICF (6 weeks if the previous chemotherapy included nitrosoureas or mitomycin)
* Prior radiotherapy to >25% of bone marrow
* Prior exposure to MAC-321

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer